CLINICAL TRIAL: NCT00205894
Title: Multicenter Feasibility Study of the Bion for Occipital Nerve Stimulation for Treatment of Chronic Headaches
Brief Title: Occipital Nerve Stimulation to Treat Chronic Headaches
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Pam Phongpharnich, Sr. Clinical Research Associate, Boston Scientific
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-B-003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-08

CONDITIONS: Headache Disorders
Keywords: Headache; Chronic headache; Migraine; Pain; Cluster headache
MeSH Terms: conditions — Headache Disorders; Headache; Migraine Disorders; Pain; Cluster Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: bion microstimulator

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a implantable device, called the bion(R), in the treatment of chronic headache. The bion microstimulator is placed underneath the skin next to the greater occipital nerve. The bion microstimulator then stimulates the nerve by generating small amounts of electrical current.

DETAILED DESCRIPTION:
Chronic migraine and chronic cluster headaches are among the most disabling medical illnesses, inflicting severe functional impairment. These headache subtypes are particularly resistant to current treatment modalities, with the majority of chronic migraine patients continuing to experience frequent or near-daily headaches despite aggressive, multidisciplinary, and multimodal therapy. The refractory nature of these illnesses and the level of devastation they inflict on the lives of their victims has motivated the pursuit of novel treatment approaches.

Direct stimulation of the greater occipital nerve has been shown to alleviate the symptoms of chronic migraine and chronic cluster headaches in a small number of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed with chronic migraine, probable chronic migraine, and/or chronic cluster headache according to the 2004 IHS Classification Criteria (2nd ed.) or be diagnosed with migraine with or without aura
2. Be 18 years of age or older
3. Be willing and able to follow all study-related procedures during the course of the study;
4. Have exhibited refractoriness to two acute medication regimens and two prophylactic medications from two separate preventative classes.

Exclusion Criteria:

1. Have received a botulinum toxin (botox) injection for treatment of headache within the last 90 days;
2. Have previously undergone destructive ganglionectomy affecting C2/C3 occipital and/or trigeminal distribution or have an occipital blockade currently in effect;
3. Have had a previous surgery in the intended implant area;
4. Have Arnold-Chiari malformation;
5. Have participated within the last 30 days or plan to participate within the next 4 months in a device or drug trial;
6. Be pregnant or planning on becoming pregnant during the study period;
7. Have an implanted electrical device (e.g., pacemaker, spinal cord stimulator) that may interfere with this therapy; and
8. Currently require, or be likely to require, MRI or diathermy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-01; Primary Completion 2006-10 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary safety measure is the incidence of major complications, defined as device or procedure related major adverse events that require medical and surgical intervention.
The primary efficacy measure is a significant reduction in the frequency, severity or duration of the headaches from the preoperative to the three-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: David Dodick, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Scottsdale, Arizona
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan

REFERENCES:
- [Derived] Trentman TL, Rosenfeld DM, Vargas BB, Schwedt TJ, Zimmerman RS, Dodick DW. Greater occipital nerve stimulation via the Bion microstimulator: implantation technique and stimulation parameters. Clinical trial: NCT00205894. Pain Physician. 2009 May-Jun;12(3):621-8. PMID 19461827